CLINICAL TRIAL: NCT02187263
Title: DZHK TranslatiOnal Registry for CardiomyopatHies Deutsches Zentrum für Herz- Und Kreislauf-Forschung (DZHK)
Brief Title: German Centre for Cardiovascular Research Cardiomyopathy Register
Acronym: TORCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Kerckhoff Klinik (Other); University Hospital Goettingen (Other); University of Hamburg-Eppendorf (Other); University of Kiel (Other); University of Luebeck (Other); Mainz University (Other); University Medical Centre Mannheim (Unknown); Ludwig-Maximilians - University of Munich (Other); Medical University of Hannover (Other); Department for Community Medicine, University Medicine Greifswald (Unknown); Goethe University (Other); Charite University, Berlin, Germany (Other); University Hospital Greifswald (Other); German Heart Institute (Other); ISAR Klinikum Munich (Industry)
Responsible Party: Sponsor
Other Study IDs: DZHK TORCH 001
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Acute Myocarditis; Dilated Cardiomyopathies; Hypertrophic Cardiomyopathies; Left Ventricular Myocardial Noncompaction Cardiomyopathy; Arrhythmogenic Right Ventricular Cardiomyopathies; Amyloidosis
Keywords: hereditary cardiomyopathy,; inflammatory cardiomyopathy,; registry,; biomaterial,; clinical trial; Patients
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — EDTA, serum, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- hereditary DCM
- inflammatory DCM
- LVNC
- HCM
- ARVC
- acute myocarditis

SUMMARY:
This is a joint project by Heidelberg University and Greifswald University.

Our objective is to establish an unique national multi-center registry and biobank of well phenotyped patients with non-ischemic cardiomyopathies (CMP) including in depth clinical, molecular and omics-based phenotyping to serve as:

1. central hub for clinical outcome studies.
2. joint resource for diagnostic and therapeutic trials.
3. common biomaterial bank.
4. resource for detailed molecular analyses on patients' biomaterials and patient specific model systems.

DETAILED DESCRIPTION:
The following basic research projects, called modules, will be tied to and rely on the recruitment of CMP patients and the infrastructure provided by TORCH:

* Well phenotyped patients will be the starting point for comprehensive next-generation genotyping, leading to advanced estimates of genotype-phenotype relationship and its clinical impact.
* Functional analysis of novel genomic loci and their related molecular pathways will be based on our established in-vitro (e.g. iPS cells, yeast two hybrid) and in-vivo (e.g. zebrafish and mice) model systems.
* The integrated analysis of viral load and replication, inflammation, genotype and clinical variables will define risk variables for inflammatory and hereditary CMP.
* By longitudinal follow-up of patients, the role of genetic, epigenetic, metabolic, molecular biomarkers and histopathology for diagnosis and out-come prediction will be defined on a national level.

The registry will also facilitate investigator initiated clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary non-ischemic cardiomyopathies including hereditary and inflammatory dilated cardiomyopathy, left ventricular non-compaction cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, and acute myocarditis.

Exclusion Criteria:

* Preexisting other cardiac diseases such as significant valvular, ischemic or pericardial disease; Severe arterial hypertension; Primary pulmonary artery hypertension; Chronic advanced disorders; History of treatment with cardiotoxic agents and chest radiation; Drug and alcohol abuse; Patients <18 and >79 years of age; Life expectancy less than 1 year due to non-cardiac comorbidity

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hereditary and inflammatory cardiomyopathies
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Time to Disease Progression | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugo A Katus, MD, Study Chair — Heidelberg University; Wolfgang Hoffmann, MD, Study Chair — Department for Community Medicine, University Medicine Greifswald
Locations (1):
- University of Heidelberg, Heidelberg, Germany